CLINICAL TRIAL: NCT06038292
Title: The Relationship Between Rheumatoid Arthritis and Osteoporosis and Factors Contributing to This Connection
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Felopateer Talaat Sedhom, felopateer talaat, Assiut University
Other Study IDs: RA&OP Relationship
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: RA & OP Relationship
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: DXA Scan — DEXA (dual x-ray absorptiometry) Scans which measure bone density (thickness and strength of bones) by passing a high and low energy x-ray beam (a form of ionizing radiation) through the body, usually in the hip, the spine and the bones of the hands and can easily diagnose osteoporosis.

SUMMARY:
This study aims to explore the association between RA and osteoporosis and highlight the risk factors that RA patients have that may cause or affect osteoporosis progress.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an autoimmune chronic connective tissue disease that produces persistent systemic inflammation, with joint inflammation leading to function loss and joint destruction. It can finally lead to some serious systematic disorders, such as cardiovascular, pulmonary, skeletal, and psychological disorders.

One of the most severe comorbidities of RA is osteoporosis (OP), which is a chronic metabolic skeletal disease leading to an increased risk of low trauma fracture, and many factors can play a role in increasing this association including treating RA patients with glucocorticoid over a long duration, chronic joints inflammation, calcium malabsorption, age of the patients, and genetics.

Osteoporosis is characterized by microarchitectural deterioration of bone tissue and low bone mass. The most commonly used measurement for OP is bone mineral density (BMD) and DEXA (dual x-ray absorptiometry) Scans.

Osteoporosis can result in devastating physical, psychosocial, and economic consequences. Still, it is often overlooked and undertreated, in large part because it is clinically silent; there are no symptoms before a fracture occurs.

Epidemiological studies indicate that about 60-80% of RA patients have a comorbidity of OP.

These two kinds of complex diseases may share some common genetic mechanisms and biological processes. For example, proinflammatory cytokines including TNF-α, IL-17, IL-6, and IL-1 have been reported to be closely associated with OP, and they also play important roles in the development of RA. Also, the inflammation in the joints increases bone absorption and makes RA patients susceptible to bone loss and osteoporosis development.

One of the primary drugs recommended for the treatment of RA is a corticosteroid, glucocorticoid (GC). Both systemic corticosteroid and intraarticular corticosteroid are proven to be risk factors for developing secondary osteoporosis and osteoporotic fracture. The risk increases with the long duration of use and using a high dose. Longer duration and severity of RA were also indicated as independent risk factors for vertebral fractures. The American College of Rheumatology (ACR) recommended increasing the awareness of RA patients about BMD and getting DXA done for identifying a patient at risk of osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 years old classified as rheumatoid arthritis based on ACR/EULAR 2010 Classification criteria.

Exclusion Criteria:

* Patients with other clinical conditions that causes secondary osteoporosis as Diabetes Mellitus, renal, liver diseases, thyroid and parathyroid disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient more than 18 years old classified as rheumatoid arthritis based on ACR/EULAR 2010 Classification criteria
  * Patients with other clinical conditions that causes secondary osteoporosis as Diabetes Mellitus, renal, liver diseases, thyroid and parathyroid disorder excluded because of probability of these disease to be a reason of osteoporosis.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with Rheumatoid Arthritis who have Osteoporosis. | baseline
  to explore the association between RA and osteoporosis and highlight the risk factors that RA patients have that may cause or affect osteoporosis progress by measuring the percentage of patents with RA who have osteoporosis.

SECONDARY OUTCOMES:
Correlation between age, disease duration, disease activity, and treatment with osteoporosis | baseline
  Correlation between age, disease duration, disease activity, and treatment with osteoporosis

REFERENCES:
- See also: Bone mineral density in patients with rheumatoid arthritis: relation between disease severity and low bone mineral density — https://ard.bmj.com/content/63/12/1576
- See also: IL-26 Is Overexpressed in Rheumatoid Arthritis and Induces Proinflammatory Cytokine Production and Th17 Cell Generation — https://journals.plos.org/plosbiology/article?id=10.1371/journal.pbio.1001395
- See also: Rheumatoid arthritis in adults: management — http://www.nice.org.uk/guidance/cg79